CLINICAL TRIAL: NCT04074213
Title: Clozapine and Haematologic Malignancies: an Observational and Retrospective Study Using the WHO Pharmacovigilance Database
Brief Title: Clozapine and Haematologic Malignancies: Observational and Retrospective Study Using the WHO Pharmacovigilance Database
Acronym: CLOZARIX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 19-916
Record Dates: First submitted 2019-08-19; First posted 2019-08-30 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma; Leukemia
MeSH Terms: conditions — Lymphoma; Leukemia | interventions — Clozapine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Haematologic malignancies with clozapine: Cases reported in the World Health Organization (WHO) database of patients treated by Clozapine, with a chronology compatible with the drug toxicity
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Clozapine — Clozapine treatment
  Other Names: Clozapine treatment

SUMMARY:
Clozapine may lead to various adverse reactions, including neutropenia and agranulocytosis. This study investigates reports of lymphoma and leukaemias for clozapine in the World Health Organization's (WHO) global database of individual safety case reports (VigiBase).

DETAILED DESCRIPTION:
Clozapine is responsible of a wide range of adverse side effects.The investigators use VigiBase, the World Health Organization (WHO) database of individual safety case reports, to identify cases of haematologic malignancies following treatment with clozapine.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 03/05/2019
* Adverse events reported were including the MedDRA terms: Malignant Lymphoma (SMQ), Leukaemia (HLGT)
* Patients treated with at least one liable antipsychotic drug (ATC class N05A)

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with at least one liable antipsychotic drug (ATC class N05A)
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between clozapine and haematologic malignancies using a disproportionality analysis in Individual Case Reports involving at least one liable antipsychotic drug in Vigibase®. | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2019 ]
  Study the correlation between clozapine and haematologic malignancies by comparing the proportion of Individual Case Reports (ICSRs) of hematologic malignancies with liable clozapine with the proportion of ICSRs of hematologic malignancies with at least one liable antipsychotic.

SECONDARY OUTCOMES:
investigate a potential dose-dependent effect | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2019 ]
  To investigate a potential dose-dependent effect, we will collect the clozapine daily dose from all clozapine ICSRs. In ICSRs with liable clozapine, the clozapine daily dose in mg will be divided into quartiles. A disproportionality analysis will be performed to evaluate the effect of the clozapine daily dose on the reporting of lymphomas and leukaemia. A significant difference of proportion of reports of haematologic malignancies between each quartile will be researched.
Description of the clinical features of clozapine-related haematologic malignancies | Case reported in the World Health Organization (WHO) of individual safety case reports to March 2019 ]
  Description of the clinical features (mean age, sex ratio, time to onset, daily dose) of clozapine-related haematologic malignancies according to the main clinical subtypes

CONTACTS AND LOCATIONS:
Overall Officials: Basile Chrétien, PharmD, MSc, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No